CLINICAL TRIAL: NCT05844488
Title: DIGITAL Biomarker: Blood Based Biomarkers in the Primary Care Setting for Timely and Accurate Diagnosis of Alzheimer's Disease
Brief Title: DIGITAL Biomarker: Blood Based Biomarkers in the Primary Care Setting for Alzheimer's Disease
Acronym: DIGITAL
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Davos Alzheimer's Collaborative (Unknown); Regenstrief Institute, Inc. (Other)
Responsible Party: Principal Investigator, Deanna Willis, Principal Investigator, Indiana University
Other Study IDs: 15289
Record Dates: First submitted 2023-04-14; First posted 2023-05-06 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Blood based biomarker group: Subjects who consent to having a blood based biomarker performed
  Interventions: Device: PrecivityAD

INTERVENTIONS:
Device: PrecivityAD — Measure risk for amyloid plaques in the brain and will include a test for certain genetic variants (specifically, ApoE proteins in the blood revealing APOE genotype) known to be associated with Alzheimer's disease.

SUMMARY:
The primary objective of this study is to evaluate the feasibility of implementing blood-based biomarker testing for amyloid positivity designed to aid the early detection of Alzheimer's Disease and Related Dementia (ADRD) in patients 65+ including the rate that patients and providers follow up abnormal blood-based biomarker testing.

DETAILED DESCRIPTION:
This study is conducted to evaluate whether a new approach to screening patients for cognitive decline in primary care practices helps with earlier detection of Alzheimer's Disease. As part of the study, the provider subjects will receive training about the PrecivityAD blood biomarker test offered by C2N Diagnostics. They will be able to order the PrecivityAD test for possible Alzheimer's disease if their patient has an abnormal screening for cognitive impairment and consents to this study. Patient subjects will have their blood drawn (1 teaspoon) for the PrecivityAD blood test and will be asked to complete a surveys before and after the blood drawn. They will receive follow up phone calls within 1 to 4 weeks after they discuss the results of their blood test with their primary care.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 65 years of age
* Any gender
* Is an established or new patient at one of the 6 participating IUHP PC sites
* Is able to provide informed consent (research portion only for the biomarker consent) or has a Legally Authorized Representative (LAR) who can provide informed consent
* Has a "red" DCA screening in the last 12 months (a score of 0 or 1 out of 5)

Exclusion Criteria:

* Patients who do not complete a DCA screening for any reason
* Existing diagnosis of dementia documented in their medical record based on ICD-10 codes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: * Patients who do not complete a DCA screening for any reason
  * Existing diagnosis of dementia documented in their medical record based on ICD-10 codes
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Patients who are willing to have Blood Based Biomarkers Performed | Mar 31, 2023 to May 31, 2023
  Evaluate the feasibility and acceptability of implementing blood-based biomarker testing for Alzhiemer's Disease and Related Dementia in primary care practices

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health Physicians Primary Care, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Identifiable individual participant data will not be shared with other researchers.